CLINICAL TRIAL: NCT07163091
Title: Bracing After Ankle Fracture (BAF): a Randomised Multicenter Non-inferiority Trial Comparing Ankle Stirrups to Walkers on Pain, Function and Social Interaction for Adults After Ankle Fracture - Study Protocol
Brief Title: Bracing After Ankle Fracture
Acronym: BAF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Randers Regional Hospital (Other); Aarhus University Hospital (Other); Viborg Regional Hospital (Other); Hospital of Southern Jutland, Aabenraa, Denmark (Unknown); Slagelse Hospital (Other); Bispebjerg Hospital (Other); Hvidovre University Hospital (Other); Herlev Hospital (Other); National Hospital of the Faroe Islands (Other Government); Hospital of South West Jutland, Esbjerg, Denmark (Unknown); Køge Hospital, Denmark (Unknown); Sygehus Lillebaelt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OP_2497/OT_0001; 10.46540/4308-00191B (Other Grant/Funding Number: Independent research fund Denmark)
Record Dates: First submitted 2025-08-20; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Ankle Fracture; Rehabilitation; Recovery
Keywords: ankle fracture; Brace; walker; ankle stirrup; intervention; RCT
MeSH Terms: conditions — Ankle Fractures | interventions — Walkers

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The data collection is blinded at baseline assessment for the local project managers. The researchers will be blinded to treatment allocation until reporting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot ankel brace (walker) (Active Comparator): Walker: immobilisation during use
  Interventions: Other: Foot-ankel brace (walker)
- Ankel stirrup (Experimental): Ankel stirrup: active ankel dorsal and plantar flextion during use
  Interventions: Other: ankel stirrup

INTERVENTIONS:
Other: ankel stirrup — Ankel stirrups are a patient preferred ankel brace that allow active ankle dorsal and plantar flexion during weightbearing while maintaining lateral stability.
  Arms: Ankel stirrup
Other: Foot-ankel brace (walker) — Walkers immobilise and stabilise the ankle during weightbearing.
  Arms: foot ankel brace (walker)

SUMMARY:
Ankle fractures are common, debilitating and usually treated with immobilisation using a foot-ankle brace (walker). Emerging evidence suggests that a less restrictive brace may reduce recovery time without increasing the risk of complications, and patients tend to prefer ankle stirrups. However, evidence supporting their non-inferiority remains limited and inconclusive. Thus, the aim is assess if an ankle stirrup is non-inferior to a standard walker in reducing pain and function measured by the Manchester-Oxford Foot Questionnaire (MOXFQ) three months after ankle fracture. The hypothesis is that ankel stirrups align better with patients preferenes for less immobilising braces and offer sufficient stability while the fracture heals. Secondarily it may lead to faster recovery of function, return to work and reduced cost. The sample size of a maximum of 1400 patients allow us to assess non-inferiority in age and sex specific subgroups and treatment (surgical or non-sugical). Non-inferiority will be assessed in a pragmatic, multicenter, randomised controlled trial involving Scandinavian orthopedic departments.

DETAILED DESCRIPTION:
Ankle fractures are the third most occuring fracture. After an ankle fracture, patients experience reduced ankle function and pain [3]. Also, evidence with moderate to high risk of bias indicate that immobilisation prolong patients recovery. However, high quality evidence are necessary for finite conclusions.

In Scandinavia, foot-ankle braces (walkers) are used to immobilise the fracture while healing. Even though patients acknowledge the need for immobilisation, a qualitative study of ten patients found that patients experienced difficulties in adhering to the recommendation of immobilisation after ankle fracture. A randomised controlled trial (RCT) by Smeeing et al. 2020 found that braces and elastic bands that allow more ankle movement than walkers did not lead to poorer functional outcomes (p=0.56), but may lead to a faster return to work (p = 0.02) without increased complications (p=0.63). The RCT was terminated when half the sample had been included, thus questioning the statistical power of the findings. Based on patient interviews completed during trial preparations we learned that patients preferred ankle stirrups as they allowed movement during use. The same patients also expressed an aversion to the walker, while being hesitant that ankle-supporting elastic bandages provided sufficient support.

Compared to the walker, ankle stirrups may better align with patient preferences while remaining non-inferior in restoring ankle-related outcomes such as pain and function.

Patients will be included in the orthopedic outpatient departments and randomised to a walker or an ankle stirrup. Randomisation will be in blocks to ensure that surgically and non-surgically patients are evenly distributed between groups and that each center will have an equal amount of intervention and control patients. Weightbearing will be unrestricted in both groups so the difference will be the brace (ankel stirrup or walker). Other variation will be a reflection of usual practice. The primary outcome is a validated score including pain, function and social interaction 12 weeks after ankel fracture. The sample size is calculated to 140 patients per each of six subgroups (males 18-39, females 18-39, males 40-59, females 40-59, males 60+, females 60+) randomisation stop when the smallest subgroup (females 18-39 years) reaches 140 or a maximum of 1400 has been included. Patients have been involved in designing the trial and a former ankle fracture patient serves a member of the steering committee.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Surgically or non-surgically treated ankle fracture

Exclusion Criteria:

* Pathological fractures
* Inadequacy to read or speak danish
* Open fractures
* Prolonged need for immobilisation (e.g. non-union or insufficient wound healing)
* Inability to adhere to trial procedures (e.g. neuropathy or severe psychiatric disorder)
* Restricted weightbearing
* Uninterest in participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Index score (0-100) of the Manchester-Oxford Foot Questionnaire (MOXFQ) | Measured as the change from baseline and after 6 and 12 weeks
  The index score of the Manchester-Oxford Foot Questionnaire (MOXFQ) three months after randomisation is chosen as the primary outcome. Patients prefer MOXFQ, and it is a valid and reliable self-administered 16-item patient-reported outcome (PRO) divided into three dimensions (walking/standing seven items, pain five items and social interaction four items). MOXFQ will be summarised as an index score covering the most important dimensions patients indicated after ankle fracture (e.g. pain, function and social interaction). Response options consist of a 5-point Likert scale ranging from zero to four. The MOXFQ index score will be calculated by summing the raw scores of the 16 items of the MOXFQ to a index score ranging from a minimum of 0 to a maximum of 100, where 100 represents the most severe health state.

SECONDARY OUTCOMES:
Physical activity | Measured as the change from baseline and after 6 and 12 weeks
  The short-form International Physical Activity Questionnaire (IPAQ-SF) measure physical activity in five domains, including work-related physical activity, transportation, housework, leisure time and time spent sitting. Patients will be grouped into low, moderate and high physical activity levels depending on activities and time spent doing these activities.
Health-related Quality Of Life (HRQOL) | Measured as the change from baseline and after 6 and 12 weeks
  HRQOL will be measured using the EuroQol five-dimension five-level questionnaire (ed-5d-5l)
Ankle dorsiflexion | Measured as the change from baseline and after 6 and 12 weeks
  is measured using the knee-to-wall test, which measures ankle mobility in degrees of motion in standing.
Ankle strength | Measured as the change from baseline and after 6 and 12 weeks
  is measured using the heel rise test. Patients perform as many single-leg heel raises at a cadence of one per second until fatigue or a maximum of 50 is reached. The test is performed on both legs, and normal function is recovered if the difference in heel raises between legs is 10% or less.
Hospital costs | Measured as the total cost from baseline and after 12 weeks
  Hospital Costs will be measured from a hospital perspective with a time horizon of three months and include cost of procedures and in-hospital activities.
Return to work | From fracture and until date of return to work.
  Will be measured by asking patients what date they returned to work (full-time and part-time). Information on work-related physical requirements (e.g., blue-collar or white-collar workers) and usual employment status (e.g., retiree, unemployed, working) will also be collected.
Index score (0-100) of the Manchester-Oxford Foot Questionnaire (MOXFQ) in subgroups | Measured as the change from baseline after 6 and 12 weeks.
  The index score of the Manchester-Oxford Foot Questionnaire (MOXFQ) three months after randomisation is chosen as the primary outcome. Patients prefer MOXFQ, and it is a valid and reliable self-administered 16-item patient-reported outcome (PRO) divided into three dimensions (walking/standing seven items, pain five items and social interaction four items). MOXFQ will be summarised as an index score covering the most important dimensions patients indicated after ankle fracture (e.g. pain, function and social interaction). Response options consist of a 5-point Likert scale ranging from zero to four. The MOXFQ index score will be calculated by summing the raw scores of the 16 items of the MOXFQ to a index score ranging from a minimum of 0 to a maximum of 100, where 100 represents the most severe health state and analysed in subgroups: males 18-39, females 18-39, males 40-59, females 40-59, males 60+, females 60+ and in treatment groups (surgical and non-surgical)
Adverse Events (AE) and Serious Adverse Events (SAE) | Safety reporting for each patient will begin at baseline and after 6 and twelve weeks
  Adverse events are undesirable experiences that may occur during brace use as: i) skin irritation, blisters, or pressure sores due to poor fit, friction, or prolonged use, ii) swelling or increased edema, iii) pain or discomfort resulting from tightness, misalignment, or mechanical pressure, iv) delayed fracture healing due to excessive joint movement, v) Muscle atrophy or joint stiffness from immobilization, vi) reduced range of motion (ROM) and vii) removal of material (e.g., screws) due to discomfort or healing complications. Serious adverse events are complications requiring hospitalisation, surgical intervention, or posing a significant risk to the patient as i) death (e.g., an unexpected cardiac event occurring during the study period) ii) hospitalisation due to falls resulting from brace-related instability, iii) wound infection requiring inpatient treatment, potentially related to brace-induced i

OTHER OUTCOMES:
The index score of the Manchester-Oxford Foot Questionnaire (MOXFQ) | Change from baseline to 6 and 12 months follow-up
  The index score of the Manchester-Oxford Foot Questionnaire (MOXFQ) three months after randomisation is chosen as the primary outcome. Patients prefer MOXFQ, and it is a valid and reliable self-administered 16-item patient-reported outcome (PRO) divided into three dimensions (walking/standing seven items, pain five items and social interaction four items). MOXFQ will be summarised as an index score covering the most important dimensions patients indicated after ankle fracture (e.g. pain, function and social interaction). Response options consist of a 5-point Likert scale ranging from zero to four. The MOXFQ index score will be calculated by summing the raw scores of the 16 items of the MOXFQ to a index score ranging from a minimum of 0 to a maximum of 100, where 100 represents the most severe health state.
Physical activity long term | Change from baseline and after 6 and 12 months
  Physical activity will be measured in longer term using the short-form International Physical Activity Questionnaire (IPAQ-SF) and grouping patients into low, moderate and high physical activity levels.
Health-related Quality Of Life (HRQOL) long term | Baseline and after 6 and 12 months
  Long term Health-related Quality Of Life (HRQOL) will be measured using the EuroQol five-dimension five-level questionnaire (ed-5d-5l)
The index score of the Manchester-Oxford Foot Questionnaire (MOXFQ) in subgroups long term | Change from baseline and after 6 and 12 months
  The index score of the Manchester-Oxford Foot Questionnaire (MOXFQ) three months after randomisation is chosen as the primary outcome. Patients prefer MOXFQ, and it is a valid and reliable self-administered 16-item patient-reported outcome (PRO) divided into three dimensions (walking/standing seven items, pain five items and social interaction four items). MOXFQ will be summarised as an index score covering the most important dimensions patients indicated after ankle fracture (e.g. pain, function and social interaction). Response options consist of a 5-point Likert scale ranging from zero to four. The MOXFQ index score will be calculated by summing the raw scores of the 16 items of the MOXFQ to a index score ranging from a minimum of 0 to a maximum of 100, where 100 represents the most severe health state and analysed in subgroups: males 18-39, females 18-39, males 40-59, females 40-59, males 60+, females 60+ and in treatment groups (surgical and non-surgical)
Incremental cost per quality adjusted life year gain | one year from baseline
  cost-utility analysis will be completed alongside the clinical trial. Reporting will be from a societal perspective and with an one year timeframe. Utility will be measured in Quality Adjusted Life Years (QALY) by assigning values from the Danish eq-5d-5l reference set (i.e. each health state is assigned a value between -0.759 to 1.000 [40]. The follow-up period will be one year (t4). Costs will be collected from national registris. These, among others, include information on admissions, out-patient visits, home care services, contacts with general practitioners and other private healthcare professionals, prescription medication and welfare subsidies due to sick leave. Hours of informal care the last week patients receive from family and friends will be collected from patients at every follow-up (t1-t4). The reported amount will be assumed stable between time points. Valuation will based on the recommendations of the Health Technology Council and reported in euros (€) using the most
carbon footprint of the trial | From baseline and after 6 and 12 weeks
  Carbon footprint of the BAF trial will be estimated by registrering activities associated with design, management and operation of the trial and summing the carbon of to estimate the overall carbon footprint (kgCO2e) using the Clinical Trial Carbon Calculator. Registered activities will be: cradle to gate estimate of ankle stirrups and foot-ankle braces, patients visits to hospital, mean of transportation to visits (car, public or bike, trial staff travel and mean of transportation to recruitments centers.
Adverse Events and Serious Adverse Events (SAE) long term | Safety reporting for each patient will begin at baseline and after 6 and 12 months
  Adverse events are undesirable experiences that may occur during brace use as: i) skin irritation, blisters, or pressure sores due to poor fit, friction, or prolonged use, ii) swelling or increased edema, iii) pain or discomfort resulting from tightness, misalignment, or mechanical pressure, iv) delayed fracture healing due to excessive joint movement, v) Muscle atrophy or joint stiffness from immobilization, vi) reduced range of motion (ROM) and vii) removal of material (e.g., screws) due to discomfort or healing complications. Serious adverse events are complications requiring hospitalisation, surgical intervention, or posing a significant risk to the patient as i) death (e.g., an unexpected cardiac event occurring during the study period) ii) hospitalisation due to falls resulting from brace-related instability, iii) wound infection requiring inpatient treatment, potentially
Physical activity | From baseline and for a minimum of 12 weeks
  A subgroup of patients will have their physical activity objectively evaluated using an accelerometer. The SENS Accelerometer is widely used and validated for young and older orthopedic patients. The accelerometer measures total accelerometer counts per day (a valid proxy for physical activity), rest time, standing time, active time (walking time, running, cycling), number of steps, movement intensity and sleep duration for four weeks. The total amount of accelerometer counts will be used to measure the level of physical activity between groups [39]. The accelerometer will be placed on the patients thigh at the day of randomization and followed for a minimum of 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Bjarke Viberg, Phd, Study Chair — Odense Universitetshospital Ortopaedkirurgisk Afdeling
Locations (16):
- Denmark (15):
  - Orthopedic Department, Hospital of Southern Jutland, Aabenraa
  - Orthopedic Department, Aalborg Universitets Hospital, Aalborg
  - Orthopedic Department, Aarhus University Hospital, Aarhus
  - Orthopedic Department, Bispebjerg Hospital, Copenhagen
  - Orthopedic Department, Hospital of South West Jutland, Esbjerg
  - Orthopedic Department, Herlev Hospital, Herlev
  - Orthopedic Department, North Zealand Hospital, Hillerød
  - Orthopedic Department, Hvidovre Hospital, Hvidovre
  - Orthopedic Department, Hospital Lillebaelt - Kolding, Kolding
  - Orthopedic Department, Zealand University Hospital - Køge, Køge
  - Orthopedic Department, Odense University Hospital, Odense
  - Orthopedic Department, Randers Hospital, Randers
  - Orthopedic Department, Slagelse Hospital, Slagelse
  - Orthopedic Department, Hospital Lillebaelt - Vejle, Vejle
  - Orthopedic Department, Viborg Hospital, Viborg
- Surgical Centre, National Hospital of the Faroe Islands, Tórshavn, Faroe Islands

IPD SHARING:
Plan to Share IPD: Yes
Access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), will be provided to anyone who wishes to access the data.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication, no end date.
Access Criteria: Any researcher, affiliated to an established institution